CLINICAL TRIAL: NCT03657264
Title: Thorough QT/QTc Study to Assess the Electrocardiographic Safety of a New Gadolinium-based Contrast Agent P03277 in Healthy Volunteers
Brief Title: Cardiac Safety Evaluation of P03277
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: GDX-44-006
Record Dates: First submitted 2018-08-31; First posted 2018-09-05 (Actual); Results first posted 2019-08-22 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers
Keywords: Gadolinium-based contrast agent; Cardiac safety; ECG; Gadopiclenol
MeSH Terms: interventions — gadopiclenol; Moxifloxacin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Williams design for a 4*4 cross over
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sequence 1 (Experimental): The sequence of administration is: P/ScD/PC/CD
  Where:
  * P = Placebo (Nacl 0.9%)
  * CD = P03277 tested at 0.1 mmol/kg
  * ScD = P03277 tested at 0.3 mmol/kg
  * PC = Positive control (moxifloxacin 400 mg - per os).
  Interventions: Drug: P03277 0.1 mmol/kg; Drug: Moxifloxacin 400mg; Drug: NaCl 0.9%; Drug: P03277 0.3 mmol/kg
- Sequence 2 (Experimental): The sequence of administration is: CD/PC/ScD/P
  Where:
  * P = Placebo (Nacl 0.9%)
  * CD = P03277 tested at 0.1 mmol/kg
  * ScD = P03277 tested at 0.3 mmol/kg
  * PC = Positive control (moxifloxacin 400 mg - per os).
  Interventions: Drug: P03277 0.1 mmol/kg; Drug: Moxifloxacin 400mg; Drug: NaCl 0.9%; Drug: P03277 0.3 mmol/kg
- Sequence 3 (Experimental): The sequence of administration is: ScD/CD/P/PC
  Where:
  * P = Placebo (Nacl 0.9%)
  * CD = P03277 tested at 0.1 mmol/kg
  * ScD = P03277 tested at 0.3 mmol/kg
  * PC = Positive control (moxifloxacin 400 mg - per os).
  Interventions: Drug: P03277 0.1 mmol/kg; Drug: Moxifloxacin 400mg; Drug: NaCl 0.9%; Drug: P03277 0.3 mmol/kg
- Sequence 4 (Experimental): The sequence of administration is: PC/P/CD/ScD
  Where:
  * P = Placebo (Nacl 0.9%)
  * CD = P03277 tested at 0.1 mmol/kg
  * ScD = P03277 tested at 0.3 mmol/kg
  * PC = Positive control (moxifloxacin 400 mg - per os).
  Interventions: Drug: P03277 0.1 mmol/kg; Drug: Moxifloxacin 400mg; Drug: NaCl 0.9%; Drug: P03277 0.3 mmol/kg

INTERVENTIONS:
Drug: P03277 0.1 mmol/kg — Single intravenous bolus injection at 2 mL/sec
  Other Names: Gadopiclenol
Drug: Moxifloxacin 400mg — One tablet per os
Drug: NaCl 0.9% — Single intravenous bolus injection at 2 mL/sec
Drug: P03277 0.3 mmol/kg — Single intravenous bolus injection at 2 mL/sec
  Other Names: Gadopiclenol

SUMMARY:
The study is a Phase I, Single center, Randomized, Cross-over Double-blind Placebo-controlled and Open-label Positive-controlled (moxifloxacin) in healthy volunteers.

The primary objective is to assess the cardiac safety after administration of P03277 to 48 healthy volunteers at dose of 0.1 mmol/kg (anticipated clinical dose) and 0.3 mmol/kg (supra-clinical dose) by evaluating the QT and QTc intervals.

DETAILED DESCRIPTION:
Each subjects will be administered with 4 products (P03277 at the 2 different doses, placebo and moxifloxacin) in a 4*4 cross over sequence balanced for first order carry over effect. Twelve subjects will be assigned to each sequence (6 males and 6 females). The volunteers will be enrolled sequentially by cohort of 8 subjects.

ECG measurements will be compared with ECG parameters collected after administration of placebo (Nacl 0.9%). The test sensitivity will be assessed using a positive control (moxifloxacin 400 mg per os) known to induce delays in QT intervals.

ELIGIBILITY:
Inclusion Criteria:

* Subject assessed as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination)
* Subject with a Body Mass Index (BMI) > 19 kg/m² and < 28 kg/m² and a weight at least of 40 kg for female and 50 kg for male and at maximum of 100 kg

Exclusion Criteria:

-

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Vanhoutte, MD, Principal Investigator — SGS Clinical Pharmacology Unit
Locations (1):
- Clinical Pharmacology unit, SGS-Life Science Service, Antwerp, Belgium

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4
Started | 12 | 12 | 12 | 12
Completed | 12 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.8 (13.5) | 41.9 (11.1) | 44.8 (11.1) | 39.8 (10.2) | 40.5 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 6 | 6 | 24
  Male | 6 | 6 | 6 | 6 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 11 | 12 | 12 | 12 | 47
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 76.3 (10.4) | 77.6 (11.1) | 75.9 (8.3) | 71.3 (9.8) | 75.3 (9.9)

OUTCOME MEASURES:

1. Primary Outcome: Change-from-baseline Mean Effect of P03277 on QT Interval Expressed as QTc According to Fridericia's Formula (∆QTcF)
Description: Each subject was monitored with a 12-lead Holter electrocardiogram (ECG). The study had to show that both 0.1 and 0.3 mmol/kg doses of P03277 do not increase the QT interval corrected by Fridericia formula (QTcF).
  The study is successful if the difference between each of the two doses of P03277 and placebo for the largest mean change from baseline for the QTcF is lower than 10 milliseconds. The baseline was defined as the mean of the 3 triplicates ECG measured within 1 hour before each product administration.
Time Frame: from 1 hour before any administration until 24 hours post-administration at the following timepoints: -1 hour, 5 min, 10 min, 20 min, 30 min, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours, 8 hours, 24 hours.
Population: The primary analysis was performed using the per protocol set which included subjects who had no major protocol deviations throughout their whole study period.
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Groups:
- P03277 0.1 mmol/kg: All subjects who received P03277 at 0.1 mmol/kg.
- P03277 0.3 mmol/kg: All subjects who received P03277 at 0.3 mmol/kg.
- Placebo: All subjects who received placebo.
Arm/Group | P03277 0.1 mmol/kg | P03277 0.3 mmol/kg | Placebo
Number analyzed (Participants) | 47 | 47 | 47
milliseconds
  5 min | 0.97 (0.88) | 5.05 (0.89) | 0.24 (0.89)
  10 min | -0.11 (0.86) | 1.34 (0.86) | -0.59 (0.86)
  20 min | -1.25 (0.88) | -1.20 (0.88) | -1.41 (0.88)
  30 min | -1.06 (0.79) | -1.26 (0.79) | -1.69 (0.79)
  1 hour | -2.72 (0.92) | -2.44 (0.92) | -2.90 (0.92)
  1.5 hours | -3.08 (0.89) | -4.64 (0.89) | -3.53 (0.89)
  2 hours | -2.08 (0.99) | -3.22 (0.99) | -2.05 (0.99)
  3 hours | 2.34 (0.98) | -1.38 (0.98) | -0.05 (0.98)
  4 hours | 0.61 (0.97) | -0.51 (0.97) | 0.33 (0.97)
  8 hours | -2.55 (1.17) | -5.59 (1.17) | -3.66 (1.17)
  24 hours | -3.18 (0.92) | -3.28 (0.92) | -3.49 (0.93)
Statistical Analysis 1: Comparison: P03277 0.1 mmol/kg vs Placebo; For the timepoint 5 min; Test type: Non-Inferiority — The upper limit of the 90% confidence interval was expected lower to the margin of 10 milliseconds for all tests; ANCOVA — p-value is not shown, as this is a non-inferiority study; Each timepoint was tested through a separate model; Least Squares Mean Difference = 0.73, 90% CI 2-sided [-1.23 to 2.69], Standard Error of Mean 1.18
Statistical Analysis 2: Comparison: P03277 0.1 mmol/kg vs Placebo; For the timepoint 10 min; Test type: Non-Inferiority — The upper limit of the 90% confidence interval was expected lower to the margin of 10 milliseconds for all tests; ANCOVA — p-value is not shown, as this is a non-inferiority study; Each timepoint was tested through a separate model; Least Squares Mean Difference = 0.48, 90% CI 2-sided [-1.32 to 2.29], Standard Error of Mean 1.09
Statistical Analysis 3: Comparison: P03277 0.1 mmol/kg vs Placebo; For the timepoint 20 min; Test type: Non-Inferiority — The upper limit of the 90% confidence interval was expected lower to the margin of 10 milliseconds for all tests; ANCOVA — p-value is not shown, as this is a non-inferiority study; Each timepoint was tested through a separate model; Least Squares Mean Difference = 0.16, 90% CI 2-sided [-1.76 to 2.08], Standard Error of Mean 1.16
Statistical Analysis 4: Comparison: P03277 0.1 mmol/kg vs Placebo; For the timepoint 30 min; Test type: Non-Inferiority — The upper limit of the 90% confidence interval was expected lower to the margin of 10 milliseconds for all tests; ANCOVA — p-value is not shown, as this is a non-inferiority study; Each timepoint was tested through a separate model; Least Squares Mean Difference = 0.63, 90% CI 2-sided [-1.09 to 2.35], Standard Error of Mean 1.04
Statistical Analysis 5: Comparison: P03277 0.1 mmol/kg vs Placebo; For the timepoint 1 hour; Test type: Non-Inferiority — The upper limit of the 90% confidence interval was expected lower to the margin of 10 milliseconds for all tests; ANCOVA — p-value is not shown, as this is a non-inferiority study; Each timepoint was tested through a separate model; Least Squares Mean Difference = 0.18, 90% CI 2-sided [-1.88 to 2.25], Standard Error of Mean 1.25
Statistical Analysis 6: Comparison: P03277 0.1 mmol/kg vs Placebo; For the timepoint 1.5 hours; Test type: Non-Inferiority — The upper limit of the 90% confidence interval was expected lower to the margin of 10 milliseconds for all tests; ANCOVA — p-value is not shown, as this is a non-inferiority study; Each timepoint was tested through a separate model; Least Squares Mean Difference = 0.45, 90% CI 2-sided [-1.47 to 2.37], Standard Error of Mean 1.16
Statistical Analysis 7: Comparison: P03277 0.1 mmol/kg vs Placebo; For the timepoint 2 hours; Test type: Non-Inferiority — The upper limit of the 90% confidence interval was expected lower to the margin of 10 milliseconds for all tests; ANCOVA — p-value is not shown, as this is a non-inferiority study; Each timepoint was tested through a separate model; Least Squares Mean Difference = -0.03, 90% CI 2-sided [-1.99 to 1.92], Standard Error of Mean 1.18
Statistical Analysis 8: Comparison: P03277 0.1 mmol/kg vs Placebo; For the timepoint 3 hours; Test type: Non-Inferiority — The upper limit of the 90% confidence interval was expected lower to the margin of 10 milliseconds for all tests; ANCOVA — p-value is not shown, as this is a non-inferiority study; Each timepoint was tested through a separate model; Least Squares Mean Difference = 2.39, 90% CI 2-sided [0.35 to 4.43], Standard Error of Mean 1.23
Statistical Analysis 9: Comparison: P03277 0.1 mmol/kg vs Placebo; For the timepoint 4 hours; Test type: Non-Inferiority — The upper limit of the 90% confidence interval was expected lower to the margin of 10 milliseconds for all tests; ANCOVA — p-value is not shown, as this is a non-inferiority study; Each timepoint was tested through a separate model; Least Squares Mean Difference = 0.27, 90% CI 2-sided [-1.57 to 2.12], Standard Error of Mean 1.11
Statistical Analysis 10: Comparison: P03277 0.1 mmol/kg vs Placebo; For the timepoint 8 hours; Test type: Non-Inferiority — The upper limit of the 90% confidence interval was expected lower to the margin of 10 milliseconds for all tests; ANCOVA — p-value is not shown, as this is a non-inferiority study; Each timepoint was tested through a separate model; Least Squares Mean Difference = 1.11, 90% CI 2-sided [-1.15 to 3.37], Standard Error of Mean 1.36
Statistical Analysis 11: Comparison: P03277 0.1 mmol/kg vs Placebo; For the timepoint 24 hours; Test type: Non-Inferiority — The upper limit of the 90% confidence interval was expected lower to the margin of 10 milliseconds for all tests; ANCOVA — p-value is not shown, as this is a non-inferiority study; Each timepoint was tested through a separate model; Least Squares Mean Difference = 0.31, 90% CI 2-sided [-1.52 to 2.14], Standard Error of Mean 1.10
Statistical Analysis 12: Comparison: P03277 0.3 mmol/kg vs Placebo; For the timepoint 5 min; Test type: Non-Inferiority — The upper limit of the 90% confidence interval was expected lower to the margin of 10 milliseconds for all tests; ANCOVA — p-value is not shown, as this is a non-inferiority study; Each timepoint was tested through a separate model; Least Squares Mean Difference = 4.81, 90% CI 2-sided [2.84 to 6.78], Standard Error of Mean 1.19
Statistical Analysis 13: Comparison: P03277 0.3 mmol/kg vs Placebo; For the timepoint 10 min; Test type: Non-Inferiority — The upper limit of the 90% confidence interval was expected lower to the margin of 10 milliseconds for all tests; ANCOVA — p-value is not shown, as this is a non-inferiority study; Each timepoint was tested through a separate model; Least Squares Mean Difference = 1.93, 90% CI 2-sided [0.12 to 3.73], Standard Error of Mean 1.09
Statistical Analysis 14: Comparison: P03277 0.3 mmol/kg vs Placebo; For the timepoint 20 min; Test type: Non-Inferiority — The upper limit of the 90% confidence interval was expected lower to the margin of 10 milliseconds for all tests; ANCOVA — p-value is not shown, as this is a non-inferiority study; Each timepoint was tested through a separate model; Least Squares Mean Difference = 0.20, 90% CI 2-sided [-1.71 to 2.12], Standard Error of Mean 1.16
Statistical Analysis 15: Comparison: P03277 0.3 mmol/kg vs Placebo; For the timepoint 30 min; Test type: Non-Inferiority — The upper limit of the 90% confidence interval was expected lower to the margin of 10 milliseconds for all tests; ANCOVA — p-value is not shown, as this is a non-inferiority study; Each timepoint was tested through a separate model; Least Squares Mean Difference = 0.43, 90% CI 2-sided [-1.29 to 2.15], Standard Error of Mean 1.04
Statistical Analysis 16: Comparison: P03277 0.3 mmol/kg vs Placebo; For the timepoint 1 hour; Test type: Non-Inferiority — The upper limit of the 90% confidence interval was expected lower to the margin of 10 milliseconds for all tests; ANCOVA — p-value is not shown, as this is a non-inferiority study; Each timepoint was tested through a separate model; Least Squares Mean Difference = 0.47, 90% CI 2-sided [-1.60 to 2.53], Standard Error of Mean 1.25
Statistical Analysis 17: Comparison: P03277 0.3 mmol/kg vs Placebo; For the timepoint 1.5 hours; Test type: Non-Inferiority — The upper limit of the 90% confidence interval was expected lower to the margin of 10 milliseconds for all tests; ANCOVA — p-value is not shown, as this is a non-inferiority study; Each timepoint was tested through a separate model; Least Squares Mean Difference = -1.11, 90% CI 2-sided [-3.03 to 0.81], Standard Error of Mean 1.16
Statistical Analysis 18: Comparison: P03277 0.3 mmol/kg vs Placebo; For the timepoint 2 hours; Test type: Non-Inferiority — The upper limit of the 90% confidence interval was expected lower to the margin of 10 milliseconds for all tests; ANCOVA — p-value is not shown, as this is a non-inferiority study; Each timepoint was tested through a separate model; Least Squares Mean Difference = -1.17, 90% CI 2-sided [-3.13 to 0.78], Standard Error of Mean 1.18
Statistical Analysis 19: Comparison: P03277 0.3 mmol/kg vs Placebo; For the timepoint 3 hours; Test type: Non-Inferiority — The upper limit of the 90% confidence interval was expected lower to the margin of 10 milliseconds for all tests; ANCOVA — p-value is not shown, as this is a non-inferiority study; Each timepoint was tested through a separate model; Least Squares Mean Difference = -1.33, 90% CI 2-sided [-3.36 to 0.71], Standard Error of Mean 1.23
Statistical Analysis 20: Comparison: P03277 0.3 mmol/kg vs Placebo; For the timepoint 4 hours; Test type: Non-Inferiority — The upper limit of the 90% confidence interval was expected lower to the margin of 10 milliseconds for all tests; ANCOVA — p-value is not shown, as this is a non-inferiority study; Each timepoint was tested through a separate model; Least Squares Mean Difference = -0.85, 90% CI 2-sided [-2.69 to 1.00], Standard Error of Mean 1.11
Statistical Analysis 21: Comparison: P03277 0.3 mmol/kg vs Placebo; For the timepoint 8 hours; Test type: Non-Inferiority — The upper limit of the 90% confidence interval was expected lower to the margin of 10 milliseconds for all tests; ANCOVA — p-value is not shown, as this is a non-inferiority study; Each timepoint was tested through a separate model; Least Squares Mean Difference = -1.94, 90% CI 2-sided [-4.19 to 0.32], Standard Error of Mean 1.36
Statistical Analysis 22: Comparison: P03277 0.3 mmol/kg vs Placebo; For the timepoint 24 hours; Test type: Non-Inferiority — The upper limit of the 90% confidence interval was expected lower to the margin of 10 milliseconds for all tests; ANCOVA — p-value is not shown, as this is a non-inferiority study; Each timepoint was tested through a separate model; Least Squares Mean Difference = 0.21, 90% CI 2-sided [-1.62 to 2.04], Standard Error of Mean 1.11

2. Secondary Outcome: Change-from-baseline Mean Effect of Moxifloxacin on QT Interval Expressed as QTc According to Fridericia's Formula (∆QTcF)
Description: Each subject was monitored with a 12-lead Holter electrocardiogram (ECG). The assay sensitivity was assessed through this outcome. The difference between the positive control (moxifloxacin) and placebo for the largest mean change from baseline for the QTcF had to be greater than 5 milliseconds for at least one time point. The baseline was defined as the mean of the 3 triplicates ECG measured within 1 hour before each product administration.
Time Frame: from 1 hour before any administration until 4 hours post-administration at the following timepoints: -1 hour, 1 hour, 1.5 hours, 2 hours, 3 hours, 4 hours.
Population: Analysis of secondary criteria was performed using the full analysis set which included all randomized subjects.
Measure: Least Squares Mean (Standard Error); unit: milliseconds
Groups:
- Positive Control (Moxifloxacin): All subjects who received moxifloxacin.
Arm/Group | Positive Control (Moxifloxacin) | Placebo
Number analyzed (Participants) | 48 | 48
milliseconds
  1 hour | 1.73 (0.91) | -2.89 (0.91)
  1.5 hours | 6.13 (0.88) | -3.27 (0.88)
  2 hours | 8.60 (0.97) | -1.95 (0.97)
  3 hours | 10.50 (0.97) | 0.17 (0.97)
  4 hours | 11.28 (0.95) | 0.63 (0.95)
Statistical Analysis 1: Comparison: Positive Control (Moxifloxacin) vs Placebo; For the timepoint 1 hour; Test type: Superiority — The lower limit of the adjusted confidence interval was expected upper to the margin of 5 milliseconds; ANCOVA — p-value is not shown, as this is a non-inferiority study; As multiple timepoints were examined separately, the overall type I error rate needed to be adjusted; Least Squares Mean Difference = 4.62, 90% CI 2-sided [2.58 to 6.66], Standard Error of Mean 1.23
Statistical Analysis 2: Comparison: Positive Control (Moxifloxacin) vs Placebo; For the timepoint 1.5 hours; Test type: Superiority — The lower limit of the adjusted confidence interval was expected upper to the margin of 5 milliseconds; ANCOVA — p-value is not shown, as this is a non-inferiority study; As multiple timepoints were examined separately, the overall type I error rate needed to be adjusted; Least Squares Mean Difference = 9.40, 90% CI 2-sided [7.14 to 11.66], Standard Error of Mean 1.14
Statistical Analysis 3: Comparison: Positive Control (Moxifloxacin) vs Placebo; For the timepoint 2 hours; Test type: Superiority — The lower limit of the adjusted confidence interval was expected upper to the margin of 5 milliseconds; ANCOVA — p-value is not shown, as this is a non-inferiority study; As multiple timepoints were examined separately, the overall type I error rate needed to be adjusted; Least Squares Mean Difference = 10.55, 90% CI 2-sided [7.92 to 13.17], Standard Error of Mean 1.16
Statistical Analysis 4: Comparison: Positive Control (Moxifloxacin) vs Placebo; For the timepoint 3 hours; Test type: Superiority — The lower limit of the adjusted confidence interval was expected upper to the margin of 5 milliseconds; ANCOVA — p-value is not shown, as this is a non-inferiority study; As multiple timepoints were examined separately, the overall type I error rate needed to be adjusted; Least Squares Mean Difference = 10.33, 90% CI 2-sided [7.70 to 12.95], Standard Error of Mean 1.22
Statistical Analysis 5: Comparison: Positive Control (Moxifloxacin) vs Placebo; For the timepoint 4 hours; Test type: Superiority — The lower limit of the adjusted confidence interval was expected upper to the margin of 5 milliseconds; ANCOVA — p-value is not shown, as this is a non-inferiority study; As multiple timepoints were examined separately, the overall type I error rate needed to be adjusted; Least Squares Mean Difference = 10.65, 90% CI 2-sided [8.05 to 13.25], Standard Error of Mean 1.10

3. Secondary Outcome: Predicted Value of ∆∆QTc at Cmax
Description: Concentration-response relationship was investigated between ∆QTc and P03277 concentrations using a mixed model approach. Plasma concentration of P03277 was measured at the same timepoints as ECG measurements.
Time Frame: from 1 hour before any administration until 24 hours post-administration.
Measure: Number (90% Confidence Interval); unit: milliseconds
Arm/Group | P03277 0.1 mmol/kg | P03277 0.3 mmol/kg
Number analyzed (Participants) | 48 | 48
milliseconds | 0.41 [-0.08 to 0.90] | 2.23 [1.19 to 3.26]

ADVERSE EVENTS:
Time Frame: From informed consent signature until the end of the confinement period, i.e. a period ranging from 32 to 41 days.
Arm/Group | P03277 0.1 mmol/kg | P03277 0.3 mmol/kg | Positive Control (Moxifloxacin) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/48 | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/48 | 0/48 | 0/48
Other Adverse Events (participants affected / at risk) | 25/48 | 22/48 | 16/48 | 22/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P03277 0.1 mmol/kg (N=48) | P03277 0.3 mmol/kg (N=48) | Positive Control (Moxifloxacin) (N=48) | Placebo (N=48)
Application site irritation (General disorders) | 6 (7) | 7 (8) | 5 (5) | 6 (6)
Injection site haematoma (General disorders) | 4 (4) | 3 (3) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Catheter site haematoma (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Injection site rash (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Catheter site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 6 (6) | 5 (6) | 4 (4) | 4 (4)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 4 (4)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-08-31): https://cdn.clinicaltrials.gov/large-docs/64/NCT03657264/Prot_002.pdf
  • Statistical Analysis Plan (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/64/NCT03657264/SAP_003.pdf